CLINICAL TRIAL: NCT02222545
Title: A Phase 2, Uncontrolled, Three-Stage, Dose-Escalation Cohort Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, Immunogenicity, and Clinical Activity of OMS721 in Adults With Thrombotic Microangiopathies
Brief Title: Safety and Efficacy Study of OMS721 in Patients With Thrombotic Microangiopathies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Omeros Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMS721-TMA-001; 2014-001032-11 (EudraCT Number)
Expanded Access: NCT04247906 (Available)
Record Dates: First submitted 2014-08-18; First posted 2014-08-21 (Estimated); Results first posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-01

CONDITIONS: Thrombotic Microangiopathies
Keywords: TMA, aHUS, HSCT-associated TMA, TTP
MeSH Terms: conditions — Thrombotic Microangiopathies; Atypical Hemolytic Uremic Syndrome | interventions — narsoplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- OMS721 low dose (Experimental): Administration of OMS721 at a low dose
  Interventions: Biological: OMS721
- OMS721 medium dose (Experimental): Administration of OMS721 at a medium dose
  Interventions: Biological: OMS721
- OMS721 high dose (Experimental): Administration of OMS721 at a high dose
  Interventions: Biological: OMS721

INTERVENTIONS:
Biological: OMS721

SUMMARY:
The purpose of this study is to assess the safety, efficacy, pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of OMS721 in patients with thrombotic microangiopathies (TMA).

DETAILED DESCRIPTION:
This is a Phase 2, uncontrolled, 3-stage, ascending-dose-escalation study in patients with 1 of 3 forms of TMA: atypical hemolytic uremic syndrome (aHUS), thrombotic thrombocytopenia (TTP), and hematopoietic stem cell transplant - associated TMA (HSCT-associated TMA). In Stage 1 of the study, OMS721 was administered to 3 cohorts, with dose escalation by cohort to identify the optimal dosing regimen. In Stage 2, the dose selected in the first stage was administered to expanded cohorts of patients with distinct etiologies (aHUS alone in 1 cohort and TTP or HSCT-TMA in the other cohort). Patients completing Stage 2 were eligible for continued treatment in Stage 3 if they tolerated OMS721 treatment and derived clinical benefit. Enrollment in the study has been completed.

ELIGIBILITY:
Inclusion Criteria:

1. Are at least age 18 at screening (Visit 1)
2. Have a diagnosis of primary aHUS, persistent HSCT-associated TMA or TTP
3. No clinically apparent alternative explanation for thrombocytopenia and anemia

Exclusion Criteria:

1. Had eculizumab therapy within three months prior to screening
2. Have STEC-HUS
3. Have a positive direct Coombs test
4. Have an active systemic bacterial or fungal infection requiring antimicrobial therapy (prophylactic antimicrobial therapy administered as standard of care is allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-11-02 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-08-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (5):
  - Omeros Investigational Site, Duarte, California
  - Omeros Investigational Site, Rochester, Minnesota
  - Omeros Investigational Site, New York, New York
  - Omeros Investigational Site, Durham, North Carolina
  - Omeros Investigational Site, Madison, Wisconsin
- Belgium (3):
  - Omeros Investigational Site, Brussels
  - Omeros Investigational Site, Leuven
  - Omeros Investigational Site, Liège
- Omeros Investigational Site, Sofia, Bulgaria
- Omeros Investigational Site, Shatin, Hong Kong
- Omeros Investigational Site, Bergamo, Italy
- Omeros Investigational Site, Vilnius, Lithuania
- Omeros Investigational Site, Selangan, Malaysia
- Omeros Investigational Site, Christchurch, New Zealand
- Poland (4):
  - Omeros Investigational Site, Katowice
  - Omeros Investigational Site, Krakow
  - Omeros Investigational Site, Lodz
  - Omeros Investigational Site, Warsaw
- Omeros Investigational Site, Singapore, Singapore
- Taiwan (2):
  - Omeros Investigational Site, Taichung
  - Omeros Investigational Site, Taipei
- Thailand (3):
  - Omeros Investigational Site, Ban Pathumwan
  - Omeros Investigational Site, Bangkok
  - Omeros Investigational Site, Pathum Thani

REFERENCES:
- [Derived] Khaled SK, Claes K, Goh YT, Kwong YL, Leung N, Mendrek W, Nakamura R, Sathar J, Ng E, Nangia N, Whitaker S, Rambaldi A; OMS721-TMA-001 Study Group Members. Narsoplimab, a Mannan-Binding Lectin-Associated Serine Protease-2 Inhibitor, for the Treatment of Adult Hematopoietic Stem-Cell Transplantation-Associated Thrombotic Microangiopathy. J Clin Oncol. 2022 Aug 1;40(22):2447-2457. doi: 10.1200/JCO.21.02389. Epub 2022 Apr 19. PMID 35439028
- [Derived] Pugh D, O'Sullivan ED, Duthie FA, Masson P, Kavanagh D. Interventions for atypical haemolytic uraemic syndrome. Cochrane Database Syst Rev. 2021 Mar 23;3(3):CD012862. doi: 10.1002/14651858.CD012862.pub2. PMID 33783815

RESULTS

PARTICIPANT FLOW:
Groups:
- OMS721 Low Dose: Administration of OMS721 at a low dose
  OMS721
- OMS721 Medium Dose: Administration of OMS721 at a medium dose
  OMS721
- OMS721 High Dose: Administration of OMS721 at a high dose
  OMS721
Period: Overall Study
Arm/Group | OMS721 Low Dose | OMS721 Medium Dose | OMS721 High Dose
Started | 3 | 3 | 52
Completed | 2 | 3 | 27
Not Completed | 1 | 0 | 25
Not completed — Adverse Event | 1 | 0 | 2
Not completed — Death | 0 | 0 | 9
Not completed — Deaths based on Long Term Chart Review of HSCT patients | 0 | 0 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 3
Not completed — Proceeded to compassionate use of OMS721 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OMS721 Low Dose | OMS721 Medium Dose | OMS721 High Dose | Total
Number analyzed (Participants) | 3 | 3 | 52 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 1
  Between 18 and 65 years | 2 | 2 | 44 | 48
  >=65 years | 1 | 0 | 8 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (17.6) | 31.7 (18.7) | 47.7 (16.1) | 46.7 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 21 | 24
  Male | 1 | 2 | 31 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 3 | 3 | 50 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 13 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 0 | 0 | 2 | 2
  White | 2 | 3 | 35 | 40
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Assess the Safety and Tolerability of Multiple-dose Administration of OMS721 in Participants With TMA
Description: Incidence of treatment-emergent adverse events (AEs): clinically significant changes in vital signs, ECG, and laboratory tests were reported as AEs.
Time Frame: Day 1 to 37 days after end of treatment, approximately up to 31 weeks.
Population: 28 participants entered the study with a diagnosis of HSCT-TMA; all participants were in the High Dose Arm
Measure: Count of Participants; unit: Participants
Groups:
- OMS721 Low Dose: Administration ofOMS721 at a low dose OMS721
Arm/Group | OMS721 Low Dose | OMS721 Medium Dose | OMS721 High Dose
Number analyzed (Participants) | 0 | 0 | 28
Participants | 0 | 0 | 27

2. Primary Outcome: Number of Participants With HSCT-TMA Who Respond to OMS721
Description: Response defined as: Improvement in TMA laboratory markers of platelet count and lactate dehydrogenase (LDH) and improvement in clinical status
Time Frame: Day 1 to up to 2 years following the first dose of OMS721
Population: Only subjects with HSCT-TMA were analyzed; 28 subjects with HSCT were in the Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | OMS721 Low Dose | OMS721 Medium Dose | OMS721 High Dose
Number analyzed (Participants) | 0 | 0 | 28
Participants | 0 | 0 | 17

3. Secondary Outcome: Participants With HSCT-TMA Treated With OMS721: 100-day Survival
Description: Number of participants alive from the date of TMA diagnosis
Time Frame: Study Day of HSCT-TMA diagnosis to 100 days later
Population: Only participants with HSCT-TMA were analyzed; all 28 HSCT-TMA participants were in the OMS721 high dose arm
Measure: Count of Participants; unit: Participants
Arm/Group | OMS721 Low Dose | OMS721 Medium Dose | OMS721 High Dose
Number analyzed (Participants) | 0 | 0 | 28
Participants | 0 | 0 | 19

4. Secondary Outcome: Participants With HSCT-TMA Treated With OMS721: Overall Survival
Description: Survival days from the day of TMA diagnosis
Time Frame: Study Day of HSCT-TMA diagnosis to up to 2 years following first dose of OMS721
Population: Only participants with HSCT-TMA were analyzed; all 28 HSCT-TMA participants were in the OMS721 high dose arm
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | OMS721 Low Dose | OMS721 Medium Dose | OMS721 High Dose
Number analyzed (Participants) | 0 | 0 | 28
days |  |  | 274 [103 to NA] — Upper limit of 95% CI not reached due to insufficient number of participants with events.

5. Secondary Outcome: Participants With HSCT-TMA Treated With OMS721: Duration of Response
Description: Number of days from the first response date to the first relapse date
Time Frame: Study Day 1 to up to 2 years following first dose of OMS721
Population: Only participants with HSCT-TMA and responded to OMS721 were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | OMS721 Low Dose | OMS721 Medium Dose | OMS721 High Dose
Number analyzed (Participants) | 0 | 0 | 17
Days |  |  | 561 [185 to 757]

6. Secondary Outcome: Participants With HSCT-TMA Treated With OMS721: Freedom From Platelet Transfusion
Description: Number of participants with absence of platelet transfusions
Time Frame: Study Day -14 to 4 weeks following the last platelet transfusion
Population: Only participants with HSCT-TMA who were receiving platelet transfusions were analyzed; all were in the OMS721 high dose arm
Measure: Count of Participants; unit: Participants
Arm/Group | OMS721 Low Dose | OMS721 Medium Dose | OMS721 High Dose
Number analyzed (Participants) | 0 | 0 | 18
Participants |  |  | 8

7. Secondary Outcome: Participants With HSCT-TMA Treated With OMS721: Freedom From Red Blood Cell (RBC) Transfusion
Description: Number of participants with absence of RBC transfusions
Time Frame: Study Day -14 to 4 weeks following the last RBC transfusion
Population: Only participants with HSCT-TMA who were receiving RBC transfusions were analyzed; all were in the OMS721 high dose arm
Measure: Count of Participants; unit: Participants
Arm/Group | OMS721 Low Dose | OMS721 Medium Dose | OMS721 High Dose
Number analyzed (Participants) | 0 | 0 | 22
Participants |  |  | 11

8. Secondary Outcome: Participants With HSCT-TMA Treated With OMS721: Change From Baseline in Platelet Count
Description: Changes from baseline in Platelet count
Time Frame: Study Day 1 to Day 97, approximately 13 weeks
Population: Only participants with HSCT-TMA were analyzed; all were in the OMS721 high dose arm
Measure: Mean (95% Confidence Interval); unit: 10^9 cells per liter
Arm/Group | OMS721 Low Dose | OMS721 Medium Dose | OMS721 High Dose
Number analyzed (Participants) | 0 | 0 | 28
10^9 cells per liter |  |  | 29.5 [13.5 to 45.6]

9. Secondary Outcome: Participants With HSCT-TMA: Pharmacokinetics (PK) of Multiple-dose Administration of OMS721
Description: PK parameters including clearance rate
Time Frame: Pre-dose and up to 204 days post-dose
Population: PK parameters were reported for all groups combined.
Measure: Mean (Standard Deviation); unit: L/H
Groups:
- HSCT-TMA: Participants in the HSCT-TMA group
Arm/Group | HSCT-TMA
Number analyzed (Participants) | 28
L/H | 0.1422 (0.0918)

10. Secondary Outcome: Participants With HSCT-TMA (ADA)
Description: Presence of ADA response. Immunogenicity of multiple-dose administration of OMS721 in subjects with TMA
Time Frame: Pre-dose and up to 204 days post-dose
Measure: Count of Participants; unit: Participants
Groups:
- OMS721-TMA-001 HSCT-TMA High Dose: 28 participants entered the study with a diagnosis of HSCT-TMA; all participants were in the high dose arm
- OMS721-TMA -001 TTP Medium Dose: 1 Patients Incidence of Treatment-Emergent Adverse Events Leading to Study Discontinuation by System Organ Class and Preferred Term for TTP
- OMS721-TMA -001 TTP High Dose: 4 Patients Incidence of Treatment-Emergent Adverse Events Leading to Study Discontinuation by System Organ Class and Preferred Term for TTP
- OMS721-TMA-001 aHUS Low Dose: 3 Patients Incidence of Treatment-Emergent Adverse Events Leading to Study Discontinuation by System Organ Class and Preferred Term for aHUS
- OMS721-TMA-001 aHUS Medium Dose: 2 Patients Incidence of Treatment-Emergent Adverse Events Leading to Study Discontinuation by System Organ Class and Preferred Term for aHUS
- OMS721-TMA-001 aHUS High Dose: 20 Patients Incidence of Treatment-Emergent Adverse Events Leading to Study Discontinuation by System Organ Class and Preferred Term for aHUS
Arm/Group | OMS721-TMA-001 HSCT-TMA High Dose | OMS721-TMA -001 TTP Medium Dose | OMS721-TMA -001 TTP High Dose | OMS721-TMA-001 aHUS Low Dose | OMS721-TMA-001 aHUS Medium Dose | OMS721-TMA-001 aHUS High Dose
Number analyzed (Participants) | 28 | 1 | 4 | 3 | 2 | 20
Participants | 3 | 0 | 1 | 1 | 0 | 6

11. Secondary Outcome: Participants With HSCT-TMA Treated With OMS721: Change From Baseline in LDH
Description: Changes from baseline in LDH
Time Frame: Study Day 1 to Day 97, approximately 13 weeks
Population: Only participants with HSCT-TMA were analyzed; all were in the OMS721 high dose arm
Measure: Mean (95% Confidence Interval); unit: U/L
Arm/Group | OMS721 Low Dose | OMS721 Medium Dose | OMS721 High Dose
Number analyzed (Participants) | 0 | 0 | 28
U/L |  |  | -111.9 [-190.7 to -33.1]

12. Secondary Outcome: Participants With HSCT-TMA Treated With OMS721: Change From Baseline in Creatine
Description: Changes from baseline in Creatine
Time Frame: Study Day 1 to Day 97, approximately 13 weeks
Population: Only participants with HSCT-TMA were analyzed; all were in the OMS721 high dose arm
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | OMS721 Low Dose | OMS721 Medium Dose | OMS721 High Dose
Number analyzed (Participants) | 0 | 0 | 28
mg/dL |  |  | -0.18 [-0.43 to 0.07]

13. Secondary Outcome: Participants With HSCT-TMA Treated With OMS721: Change From Baseline in Haptoglobin
Description: Changes from baseline in Haptoglobin
Time Frame: Study Day 1 to Day 97, approximately 13 weeks
Population: Only participants with HSCT-TMA were analyzed; all were in the OMS721 high dose arm
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | OMS721 Low Dose | OMS721 Medium Dose | OMS721 High Dose
Number analyzed (Participants) | 0 | 0 | 27
mg/dL |  |  | 67.7 [40.2 to 95.2]

14. Secondary Outcome: Participants With HSCT-TMA Treated With OMS721: Change From Baseline in Hemoglobin
Description: Changes from baseline in Hemoglobin
Time Frame: Study Day 1 to Day 97, approximately 13 weeks
Population: Only participants with HSCT-TMA were analyzed; all were in the OMS721 high dose arm
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | OMS721 Low Dose | OMS721 Medium Dose | OMS721 High Dose
Number analyzed (Participants) | 0 | 0 | 22
g/dL |  |  | 0.38 [-0.17 to 0.92]

15. Secondary Outcome: Participants With HSCT-TMA: Pharmacokinetics (PK) of Multiple-dose Administration of OMS721
Description: PK parameters Apparent volume of the central compartment (V1)
Time Frame: Pre-dose and up to 204 days post-dose
Population: PK parameters were reported for all groups combined.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | HSCT-TMA
Number analyzed (Participants) | 28
L
  Apparent volume of the central compartment (V1) | 11.6 (3.8)
  Apparent volume of the peripheral compartment (V2) | 5.6 (3.2)

16. Secondary Outcome: Participants With HSCT-TMA: Pharmacokinetics (PK) of Multiple-dose Administration of OMS721
Description: PK parameters Concentration of OMS721 that achieves half maximum elimination rate (KM) (ug/mL)
Time Frame: Pre-dose and up to 204 days post-dose
Population: PK parameters were reported for all groups combined.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | HSCT-TMA
Number analyzed (Participants) | 28
ug/mL | 14.2 (15.2)

17. Secondary Outcome: Participants With HSCT-TMA: Pharmacodynamics (PD)
Description: PD measure is expressed as percentage inhibition of C4d to assess ex-vivo lectin pathway activation
Time Frame: Pre-dose and up to 204 days post-dose
Population: PD was analyzed only in HSCT-TMA participants
Measure: Mean (Standard Deviation); unit: Percentage
Groups:
- HSCT-TMA: 28 participants entered the study with a diagnosis of HSCT-TMA; all participants were in the high dose arm
Arm/Group | HSCT-TMA
Number analyzed (Participants) | 28
Percentage
  Baseline inhibition ex vivo lectin-mediated C4d Formation % | 26.3 (31.8)
  Maximum inhibition ex vivo lectin-mediated Cd4 Formation % | 95.9 (1.21)

ADVERSE EVENTS:
Time Frame: The Adverse Event period of time was from the date of Consent to 2 years after the first dose of study drug.
Description: AEs are assessed throughout the study up to 2 years.
Groups:
- HSCT-TMA-001 High Dose (N=28): 28 participants entered the study with a diagnosis of HSCT-TMA
- aHUS OMS721-TMA-001 Low Dose: Incidence of Treatment-Emergent Adverse Events Leading to Study Discontinuation by System Organ Class and Preferred Term reported for 3 patients with aHUS
- aHUS OMS721-TMA-001 Medium Dose: Incidence of Treatment-Emergent Adverse Events Leading to Study Discontinuation by System Organ Class and Preferred Term reported for 2 patients with aHUS
- aHUS OMS721-TMA-001 High Dose: Incidence of Treatment-Emergent Adverse Events Leading to Study Discontinuation by System Organ Class and Preferred Term reported for 20 patients with aHUS
- TTP OMS721-TMA-001 Medium Dose: Incidence of Treatment-Emergent Adverse Events Leading to Study Discontinuation by System Organ Class and Preferred Term reported by 1 patients with TTP
- TTP OMS721-TMA-001 High Dose: Incidence of Treatment-Emergent Adverse Events Leading to Study Discontinuation by System Organ Class and Preferred Term reported by 4 patients with TTP
Arm/Group | HSCT-TMA-001 High Dose (N=28) | aHUS OMS721-TMA-001 Low Dose | aHUS OMS721-TMA-001 Medium Dose | aHUS OMS721-TMA-001 High Dose | TTP OMS721-TMA-001 Medium Dose | TTP OMS721-TMA-001 High Dose
All-Cause Mortality (participants affected / at risk) | 16/28 | 0/3 | 0/2 | 3/20 | 0/1 | 0/4
Serious Adverse Events (participants affected / at risk) | 17/28 | 2/3 | 0/2 | 12/20 | 0/1 | 2/4
Other Adverse Events (participants affected / at risk) | 27/28 | 2/3 | 1/2 | 19/20 | 0/1 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HSCT-TMA-001 High Dose (N=28) (N=28) | aHUS OMS721-TMA-001 Low Dose (N=3) | aHUS OMS721-TMA-001 Medium Dose (N=2) | aHUS OMS721-TMA-001 High Dose (N=20) | TTP OMS721-TMA-001 Medium Dose (N=1) | TTP OMS721-TMA-001 High Dose (N=4)
SAE by System Organ (Infections and infestations) | 10 | 1 | 0 (0) | 7 | 0 (0) | 0
SAE by System Organ (Blood and lymphatic system disorders) | 3 | 0 | 0 | 3 | 0 | 2
SAE by System Organ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0
SAE by System Organ (Immune system disorders) | 5 | 0 | 0 | 1 | 0 | 0
SAE by System Organ (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
SAE by System Organ (Psychiatric disorders) | 3 | 0 | 0 | 1 | 0 | 0
SAE by System Organ (Nervous system disorders) | 2 | 0 | 0 | 4 | 0 | 0
SAE by System Organ (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
SAE by System Organ (Vascular disorders) | 1 | 0 | 0 | 3 | 0 | 0
SAE by System Organ (Gastrointestinal disorders) | 3 | 0 | 0 | 1 | 0 | 0
SAE by System Organ (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
SAE by System Organ (Renal and urinary disorders) | 3 | 0 | 0 | 1 | 0 | 0
SAE by System Organ (General disorders) | 2 | 2 | 0 | 1 | 0 | 0
SAE by System Organ (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
SAE by System Organ (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
SAE by System Organ (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HSCT-TMA-001 High Dose (N=28) (N=28) | aHUS OMS721-TMA-001 Low Dose (N=3) | aHUS OMS721-TMA-001 Medium Dose (N=2) | aHUS OMS721-TMA-001 High Dose (N=20) | TTP OMS721-TMA-001 Medium Dose (N=1) | TTP OMS721-TMA-001 High Dose (N=4)
AE by System Organ (Infections and infestations) | 20 | 2 | 0 | 14 | 0 | 1
AE by System Organ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 1 | 0 | 0
AE by System Organ (Blood and lymphatic system disorders) | 13 | 0 | 0 | 7 | 0 | 2
AE by System Organ (Immune system disorders) | 10 | 0 | 0 | 1 | 0 | 1
AE by System Organ (Endocrine disorders) | 2 | 0 | 0 | 0 | 0 | 0
AE by System Organ (Metabolism and nutrition disorders) | 16 | 0 | 0 | 4 | 0 | 0
AE by System Organ (Psychiatric disorders) | 6 | 0 | 0 | 1 | 0 | 0
AE by System Organ (Nervous system disorders) | 10 | 0 | 0 | 5 | 0 | 2
AE by System Organ (Eye disorders) | 2 | 1 | 0 | 1 | 0 | 1
AE by System Organ (Cardiac disorders) | 7 | 0 | 0 | 3 | 0 | 0
AE by System Organ (Vascular disorders) | 8 | 0 | 1 | 8 | 0 | 0
AE by System Organ (Respiratory, thoracic and mediastinal disorders) | 13 | 0 | 0 | 1 | 0 | 1
AE by System Organ (Gastrointestinal disorders) | 18 | 0 | 0 | 0 | 0 | 0
AE by System Organ (Hepatobiliary disorders) | 3 | 0 | 0 | 1 | 0 | 0
AE by System Organ (Skin and subcutaneous tissue disorders) | 10 | 0 | 0 | 4 | 0 | 0
AE by System Organ (Musculoskeletal and connective tissue disorders) | 12 | 0 | 0 | 3 | 0 | 0
AE by System Organ (Renal and urinary disorders) | 6 | 1 | 0 | 1 | 0 | 0
AE by System Organ (General disorders) | 18 | 2 | 0 | 5 | 0 | 0
AE by System Organ (Investigations) | 10 | 1 | 0 | 3 | 0 | 0
AE by System Organ (Injury, poisoning and procedural complications) | 6 | 1 | 0 | 3 | 0 | 0
AE by System Organ (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0
AE by System Organ (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 — Dysmenorrhoea
AE by System Organ (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 — Vertigo

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT02222545/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT02222545/SAP_001.pdf